CLINICAL TRIAL: NCT01781208
Title: Ultrasound Based Acoustic Radiation Force Impulse, Shear Wave Velocity Imaging in Pediatric Patients Undergoing Liver Biopsy
Brief Title: Ultrasound Based Acoustic Radiation Force Impulse Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jonathan R. Dillman M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00063736
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Liver Fibrosis; Liver Inflammation
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound-based Acoustic Radiation Force Imaging (Experimental): The liver was scanned using ultrasound and ultrasound-based acoustic radiation force impulse imaging technique (ARFI).
  Interventions: Device: Ultrasound-Based Acoustic Radiation Force Impulse (ARFI)

INTERVENTIONS:
Device: Ultrasound-Based Acoustic Radiation Force Impulse (ARFI) — Research scans using ultrasound-based acoustic radiation force impulse (ARFI) will image the liver non-invasively.

SUMMARY:
ARFI (Ultrasound-based Acoustic Radiation Force Impulse) will be used during ultrasound guided needle biopsy of the liver of children.

DETAILED DESCRIPTION:
A new technique based on ultrasound, known as Acoustic Radiation Force Impulse (ARFI) imaging is performed using standard approved ultrasound machines and transducers. The sound waves or impulses are generated in a different pattern and offer information on the stiffness of the tissue. This new technique will be evaluated for usefulness in diagnosing different liver conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or younger
* Scheduled to have a needle biopsy of the liver at

  1. C.S. Mott Children's Hospital or
  2. Dept. of Radiology at the Univ. of Michigan Hospital
* Scheduled to have an abdominal ultrasound to evaluate your liver (with no known liver disease)

Exclusion Criteria:

* None to list

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric patients aged 18 and younger were scheduled for a liver biopsy at a large pediatric hospital between 2012 and 2014. A total of 62 patients were recruited and enrolled. Patients and their parents gave consent/assent for the study.
Groups:
- Ultrasound-based Acoustic Radiation Force Impulse (ARFI): 62 children undergoing clinically ordered ultrasound-directed percutaneous core needle liver biopsy were included. Biopsy was performed for known or suspected (non-neoplastic) liver disease. (One child did not undergo a liver biopsy, so was ineligible and not included in the above total.)
  The patients received an additional ultrasound for research purposes that utilized a technique known as ARFI. ARFI, or Acoustic Radiation Force Impulse, uses a transducer which directs sound waves again the liver to measure the stiffness of the tissues.
Period: Overall Study
Arm/Group | Ultrasound-based Acoustic Radiation Force Impulse (ARFI)
Started | 62
Overall Study | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Children undergoing percutaneous core needle liver biopsy
Groups:
- Ultrasound-based Acoustic Radiation Force Impulse (ARFI): 62 children undergoing clinically ordered ultrasound-directed percutaneous core needle liver biopsy for known or suspected (non-neoplastic) liver disease were included in this study. Subjects were between 0-18 years of age.
Arm/Group | Ultrasound-based Acoustic Radiation Force Impulse (ARFI)
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 62
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 8.0 [0 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: ARFI/VTQ and ARFI/VTIQ Liver Shear Wave Speed vs. Liver Histologic Fibrosis Score
Description: Tissue shear wave speed is positively correlated to a material's/tissue's stiffness and can be noninvasively measured by ultrasound. The relationship between liver shear wave speed and liver histologic fibrosis score were assessed using 2 different ultrasound methods. Liver shear wave speed as obtained using 2 different ultrasound methods served as our primary outcome measures.
  Note, the histologic scoring system (Ishak) ranged from 0 to 6, where 0 = no fibrosis and 6 = cirrhosis.
Time Frame: 10 minutes
Population: 49 pediatric subjects underwent successful (diagnostic) liver ARFI/VTQ) assessment and liver histologic fibrosis scoring. 13 subjects had non-diagnostic ARFI/VTQ exams.
  48 pediatric subjects underwent successful (diagnostic) liver ARFI/VTIQ) assessment and liver histologic fibrosis scoring. 14 subjects had non-diagnostic ARFI/VTIQ exams.
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Children Undergoing Diagnostic ARFI/VTQ and Fibrosis Scoring: We measured correlation between liver shear wave speed as determined by ARFI (VTQ) and liver histologic fibrosis score.
- Children Undergoing Diagnostic ARFI/VTIQ and Fibrosis Scoring: We measured correlation between liver shear wave speed as determined by ARFI/VTIQ and liver histologic fibrosis score.
Arm/Group | Children Undergoing Diagnostic ARFI/VTQ and Fibrosis Scoring | Children Undergoing Diagnostic ARFI/VTIQ and Fibrosis Scoring
Number analyzed (Participants) | 49 | 48
m/s | 1.69 (0.42) | 2.01 (0.58)
Statistical Analysis 1: Comparison: Children Undergoing Diagnostic ARFI/VTQ and Fibrosis Scoring; Continuous data were summarized using means and standard deviations. The relationship between ARFI (VTQ) liver shear wave speed and liver histologic fibrosis score were assessed using Pearson correlation. No a priori power analysis was performed; Test type: Superiority or Other; p < 0.0001, Pearson Correlation — r=0.68, unadjusted for age, gender, and histologic inflammation
Statistical Analysis 2: Comparison: Children Undergoing Diagnostic ARFI/VTIQ and Fibrosis Scoring; Continuous data were summarized using means and standard deviations. The relationship between ARFI (VTIQ) liver shear wave speed and liver histologic fibrosis score were assessed using Pearson correlation. No a priori power analysis was performed; Test type: Superiority or Other; p < 0.0001, Pearson Correlation — r=0.73, unadjusted for age, gender, and histologic inflammation score

ADVERSE EVENTS:
Time Frame: 19 months
Description: There were no adverse events
Groups:
- All Participants: No serious or non-serious adverse events were observed during the study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No